CLINICAL TRIAL: NCT03211611
Title: Role of General Practionners in Management of Women With BRCA1/2 Mutation
Brief Title: Management of Women With BRCA1/2 Mutation
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0200
Record Dates: First submitted 2017-07-06; First posted 2017-07-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2017-07

CONDITIONS: BRCA1 Mutation; BRCA2 Mutation
Keywords: BRCA1/2 Mutation; Breast cancer; General practitionner
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with BRCA ½ mutation: Women with BRCA 1 / 2 mutation with or without cancer Age over 18
  Interventions: Behavioral: Questionnaire given to the two groups
- GP: GP of the patients with BRCA 1 / 2 mutation
  Interventions: Behavioral: Questionnaire given to the two groups

INTERVENTIONS:
Behavioral: Questionnaire given to the two groups — Questionnaire given to the two groups :
  Patients with BRCA ½ mutation GP

SUMMARY:
The aim of this study is to determine general practitionners' role in management of women with BRCA1/2 mutation.

This study will be conduct between April 2017 and December 2017 at Montpellier University Hospital on women followed-up in the department of genetics and their general practitionners (GP). Patients and their GP will be called by the investigators and questionnaire will be given to them. Questionnaire includes questions for patients and their GP. The primary endpoint was to determine the rate of GP having sufficient knowledge of the adequate management of patients with BRCA1 / 2 mutation. Adequate knowledge includes : systematic search for a family history of cancer, knowing criteria required to refer women in oncogenetic department, and the ability to respond to patients' questions. Secondary endpoint was to determine women' opinion on their GP : whether or not well managed for their BRCA 1 / 2 mutation.

DETAILED DESCRIPTION:
PURPOSE: The aim of this study is to determine general practitionners' role in management of women with BRCA1/2 mutation.

METHODS:

This study will be conduct between April 2017 and December 2017 at Montpellier University Hospital on women followed-up in the department of genetics and their general practitionners (GP). Patients and their GP will be called by the investigators and questionnaire will be given to them. Questionnaire includes questions for patients and their GP. The primary endpoint was to determine the rate of GP having sufficient knowledge of the adequate management of patients with BRCA1 / 2 mutation. Adequate knowledge includes : systematic search for a family history of cancer, knowing criteria required to refer women in oncogenetic department, and the ability to respond to patients' questions. Secondary endpoint was to determine women' opinion on their GP : whether or not well managed for their BRCA 1 / 2 mutation.

ELIGIBILITY:
Inclusion criteria

* Aged over 18
* Women
* Living in France
* Having a medical insurance

Exclusion criteria

* Men
* Dementia
* Non frenchspeaker
* Mental retardation
* Being the subject of a guardianship or tutelage measure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' group: women with BRCA 1 / 2 mutation followed-up in the department of genetics at Montpellier University Hospital.
  GP group: GP of women included in patients' group.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
The rate of GP having sufficient knowledge of the adequate management of patients with BRCA1 / 2 mutation. | 1 day
  Adequate knowledge includes : systematic search for a family history of cancer, knowing criteria required to refer women in oncogenetic department, and the ability to respond to patients' questions

SECONDARY OUTCOMES:
Women' opinion on their GP | 1 day
  Women' opinion on their GP : whether or not well managed for their BRCA 1 / 2 mutation.
  The rate of GP wanting a formation in oncogenetic

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PUJOL, PR, Study Chair — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC